CLINICAL TRIAL: NCT06060639
Title: Variation of Echocardiographic Parameters After Red Blood Cell Transfusion in Emergency Department Anemic Patients
Acronym: Trans-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A01236-39
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Age Problem; Ultrasonography
MeSH Terms: conditions — Anemia | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transfused patients (Experimental): patients receiving red blood cell transfusion
  Interventions: Diagnostic Test: transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: transthoracic echocardiography — E wave, A wave, e' and vdi measurement

SUMMARY:
The goal of this interventional study is to asses echocardiographic variations in emergency department's elderly patients receiving red blood cell transfusion. The main questions it aims to answer are :

* is there a modification of echocardiographic parameters after red blood cell transfusion ?
* which parameter is the most impacted by red blood cell transfusion ? Participants will have a transthoracic echocardiography before, just after and 15 minutes after red blood cell transfusion.

ELIGIBILITY:
Inclusion Criteria:

* patient needing red blood cell transfusion
* consent
* social protection

Exclusion Criteria:

* fluid filing over 500 mL of crystalloids
* transfusion in the last hour

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
E/A ratio modification | Base line, just after and 15 minutes after red blood cell transfusion
  E/A ratio permits to estimate left ventricle pressure

SECONDARY OUTCOMES:
E/e' ratio modification | Base line, just after and 15 minutes after red blood cell transfusion
  E/e' assesses left ventricle diastolic function
E wave deceleration time | Base line, just after and 15 minutes after red blood cell transfusion
  E wave deceleration time is a reflect of left atrium pressures
Velocity-time Integral (VTI) modification | Base line, just after and 15 minutes after red blood cell transfusion
  Aortic velocity-time integral is the reflect of cardiac output
Lung score modification | Base line, just after and 15 minutes after red blood cell transfusion
  Lung score permits to asses if extravascular water is present in lungs
New York Heart Association scale (NYHA) modification | baseline and 24 hour after red blood cells transfusion
  NYHA is a validated scale to asses patient dyspnea

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pelton WJ, McNeal DR, Goggans JK. Student dental health program of the University of Alabama in Birmingham. IV. Enrollment and utilization. Ala J Med Sci. 1971 Jul;8(3):283-7. No abstract available. PMID 5112924
- [Background] Weiss A, Beloosesky Y, Gingold-Belfer R, Leibovici-Weissman Y, Levy Y, Mulla F, Issa N, Boltin D, Koren-Morag N, Meyerovitch J, Sharon E, Schmilovitz-Weiss H. Association of Anemia with Dementia and Cognitive Decline among Community-Dwelling Elderly. Gerontology. 2022;68(12):1375-1383. doi: 10.1159/000522500. Epub 2022 Mar 22. PMID 35316810
- [Background] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Background] Peyrony O, Gamelon D, Brune R, Chauvin A, Ghazali DA, Yordanov Y, Arsicaud A, Gilleron P, Curac S, Richard MC, Feral-Pierssens AL, Villoing B, Beaune S, Goulet H, Fontaine JP, Francois A, Pirenne F. Red Blood Cell Transfusion in the Emergency Department: An Observational Cross-Sectional Multicenter Study. J Clin Med. 2021 Jun 2;10(11):2475. doi: 10.3390/jcm10112475. PMID 34199655
- [Background] Kracalik I, Mowla S, Basavaraju SV, Sapiano MRP. Transfusion-related adverse reactions: Data from the National Healthcare Safety Network Hemovigilance Module - United States, 2013-2018. Transfusion. 2021 May;61(5):1424-1434. doi: 10.1111/trf.16362. Epub 2021 Apr 20. PMID 33880771
- [Background] Roubinian N. TACO and TRALI: biology, risk factors, and prevention strategies. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):585-594. doi: 10.1182/asheducation-2018.1.585. Epub 2018 Dec 14. PMID 30570487
- [Background] Klanderman RB, Bosboom JJ, Migdady Y, Veelo DP, Geerts BF, Murphy MF, Vlaar APJ. Transfusion-associated circulatory overload-a systematic review of diagnostic biomarkers. Transfusion. 2019 Feb;59(2):795-805. doi: 10.1111/trf.15068. Epub 2018 Nov 29. PMID 30488959
- [Background] Morita T, Nakamura K, Osuga T, Yokoyama N, Morishita K, Sasaki N, Ohta H, Takiguchi M. Effect of acute volume overload on echocardiographic indices of right ventricular function and dyssynchrony assessed by use of speckle tracking echocardiography in healthy dogs. Am J Vet Res. 2019 Jan;80(1):51-60. doi: 10.2460/ajvr.80.1.51. PMID 30605034
- [Background] Bosboom JJ, Klanderman RB, Terwindt LE, Bulle EB, Wijnberge M, Eberl S, Driessen AH, Winkelman TA, Geerts BF, Veelo DP, Hollmann MW, Vlaar APJ. Autologous red blood cell transfusion does not result in a more profound increase in pulmonary capillary wedge pressure compared to saline in critically ill patients: A randomized crossover trial. Vox Sang. 2022 Aug;117(8):1035-1042. doi: 10.1111/vox.13292. Epub 2022 May 13. PMID 35560234
- [Background] Dencker M, Stagmo M. Reported normal values and weighted means for commonly used echocardiography pulsed Doppler and tissue Doppler measurements. Clin Physiol Funct Imaging. 2018 May;38(3):341-350. doi: 10.1111/cpf.12427. Epub 2017 Apr 12. PMID 28402044